CLINICAL TRIAL: NCT00624039
Title: The Effect of Cataract Extraction on the Contractility of Ciliary Muscle
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Samsung Medical Center (Other)
Responsible Party: Changwon Kee, Department of Ophthalmology, Samsung Medical Center, Seoul, Korea
Allocation: Not Applicable | Model: Single Group | Masking: Double | Purpose: Basic Science
Other Study IDs: CB2006
Record Dates: First submitted 2008-02-18; First posted 2008-02-26 (Estimated); Last update posted 2008-02-26 (Estimated); Status verified 2006-05

CONDITIONS: Presbyopia; Cataract
Keywords: presbyopia
MeSH Terms: conditions — Presbyopia; Cataract | interventions — Pilocarpine

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Other): ultrasound biomicrocopic examinations and pilocarpine instillation
  Interventions: Other: UBM with pilocarpine in presbyopia

INTERVENTIONS:
Other: UBM with pilocarpine in presbyopia — ultrasound biomicroscopic examination in both eyes 30 minutes after one drop of 2% pilocarpine hydrochloride (Ocucarpine®, Samil Pharm., Seoul, Korea) instillation before and two months after cataract surgery
  Other Names: UBM with pilocarpine

SUMMARY:
The purpose of this study is to investigate the changes in the pilocarpine-induced ciliary body movement before and after cataract extraction in order to determine the effect of lens sclerosis on the ciliary muscle contractility.

DETAILED DESCRIPTION:
The functional changes in the ciliary body in presbyopia are not only important in a study of the mechanism for presbyopia but are also a key to various procedures or devices used to restore accommodation. Therefore, it is becoming increasingly important to quantify the in vivo accommodative changes in the aging ciliary muscle with and without a lens. We are going to evaluate the changes in the pilocarpine-induced contractility of the ciliary muscle in eyes with presbyopia before and after cataract extraction using ultrasound biomicroscopy (UBM).UBM will be performed with and without instilling 2 % pilocarpine, as well as before and 2 months after cataract extraction. Images of the ciliary body will be compared visually using Adobe Photoshop 7.0.

ELIGIBILITY:
Inclusion Criteria:

* Age : same or more than 55 years
* Patients with senile cataract who are going to get cataract surgery

Exclusion Criteria:

* Age : less than 55 years
* Previous ocular disease other than cataract.

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2006-05; Primary Completion 2008-03 (Estimated); Study Completion 2008-03 (Estimated)

PRIMARY OUTCOMES:
ultrasound biomicroscopic findings (ciliary body axial length) | 2 months before and after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Changwon Kee, M.D., Study Director — Department of Ophthalmology, Samsung Medical Center, Ilwon-dong, Kangnam-gu, Seoul, 135-710, Republic of Korea. E-mail: ckee@skku.edu
Locations (1):
- Samsung Medical Center, Seoul, South Korea

REFERENCES:
- [Background] Stachs O, Martin H, Kirchhoff A, Stave J, Terwee T, Guthoff R. Monitoring accommodative ciliary muscle function using three-dimensional ultrasound. Graefes Arch Clin Exp Ophthalmol. 2002 Nov;240(11):906-12. doi: 10.1007/s00417-002-0551-2. Epub 2002 Oct 9. PMID 12486512